CLINICAL TRIAL: NCT00863018
Title: Change in Corneal Endothelium After Glaucoma Surgery; Trabeculectomy and Glaucoma Implant Surgery
Brief Title: Corneal Endothelium After Glaucoma Surgery
Status: Completed | Type: Observational
Sponsor: Chungnam National University (Other)
Responsible Party: Principal Investigator, Chang-sik Kim, professor, Chungnam National University
Other Study IDs: CNUMC-09-04
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Glaucoma; Corneal Damage; Intraocular Pressure
Keywords: Corneal endothelial cell; Specular microscopy; Glaucoma implant surgery; Ahmed glaucoma valve; Trabeculectomy
MeSH Terms: conditions — Glaucoma; Corneal Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control: Eyes with glaucoma and on anti-glaucoma medication but without glaucoma surgery
- Implant surgery: Eyes underwent Ahmed glaucoma valve implantation
- Trabeculectomy: Eyes underwent conventional trabeculectomy with mitomycin-C

SUMMARY:
The purpose of this trial is to study the change in corneal endothelial cell after glaucoma surgery, non-contact specular microscopic examination is performed for the patients who underwent glaucoma surgery; trabeculectomy and Ahmed glaucoma valve implant surgery prospectively. Change in corneal endothelial cell density, hexagonality, and coefficient of variation of cell area will be analyzed and compared to the baseline and between the types of the surgeries.

DETAILED DESCRIPTION:
To study the change in corneal endothelial cell after glaucoma surgery, non-contact specular microscopic examination is performed for the patients who underwent glaucoma surgery; trabeculectomy and Ahmed glaucoma valve implant surgery prospectively. Specular microscopy using non-contact type specular microscope (Noncon Robo SP-8000, Konan Medical Inc., Tokyo, Japan) was performed by one experienced examiner before surgery and 1, 6, 12, 18, and 24 months after surgery. All examinations were done at the center, superior, superonasal, and superotemporal area of the cornea, while the patient maintain fixation at the target in the equipment. The follow-up was stopped if serious complication requiring surgical treatment was developed or additional intraocular pressure lowering surgery is needed, and the data before the second surgery were collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need glaucoma surgery for intraocular pressure control

Exclusion Criteria:

* congenital glaucoma
* Pre-existing corneal abnormality
* lost from follow up without any ocular problem within 6 months from surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent glaucoma surgery; trabeculectomy and Ahmed glaucoma valve implant surgery
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2003-08; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in corneal endothelial cell density, hexagonality, and coefficient of variation of cell area | 1 and 2 years longitudinal follow up

SECONDARY OUTCOMES:
Clinical factors associated with the damage of corneal endothelium after glaucoma surgery | 1 and 2 years longitudinal follow up

CONTACTS AND LOCATIONS:
Overall Officials: Young-ha Lee, MD, PhD, Study Director — Research Institute for Medical Science, Chungnam National University; Chang-sik Kim, MD, PhD, Principal Investigator — Ophthalmology, College of Medicine, Chungnam National University
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

REFERENCES:
- [Derived] Lee EK, Yun YJ, Lee JE, Yim JH, Kim CS. Changes in corneal endothelial cells after Ahmed glaucoma valve implantation: 2-year follow-up. Am J Ophthalmol. 2009 Sep;148(3):361-7. doi: 10.1016/j.ajo.2009.04.016. Epub 2009 Jun 7. PMID 19505676